CLINICAL TRIAL: NCT02022501
Title: A Phase I/II, Open-label, Dose-escalating, Sequential-cohort Study Assessing the Safety, Tolerability, Pharmacokinetics and Bioactivity of a Single Intravitreal Injection of DE-120 Injectable Solution for the Treatment of Late Stage Exudative Age-related Macular Degeneration
Brief Title: A Phase I/II Safety Study of DE-120 Injectable Solution for Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35-001
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Age-Related Macular Degeneration
Keywords: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose DE-120 (Experimental): Single 20 µL intravitreal injection of Low Dose DE-120 injectable solution
  Interventions: Drug: DE-120
- Medium Dose DE-120 (Experimental): Single 20 µL intravitreal injection of Medium Dose DE-120 injectable solution
  Interventions: Drug: DE-120
- High Dose DE-120 (Experimental): Single 20 µL intravitreal injection of High Dose DE-120 injectable solution
  Interventions: Drug: DE-120

INTERVENTIONS:
Drug: DE-120

SUMMARY:
The purpose of this study is to assess the safety, tolerability, bioactivity and pharmacokinetics of three concentrations of DE-120 after a single intravitreal injection in subjects with late stage exudative age-related macular degeneration.

DETAILED DESCRIPTION:
This is an open-label, dose-escalating, sequential-cohort study of DE-120 injectable solution administered in 9, and up to 12, subjects with late stage exudative age-related macular degeneration.

Three cohorts of 3 subjects will receive a single intravitreal injection in the study eye. Subjects in Cohort 1 will receive a single intravitreal injection of Low Dose DE-120 injectable solution in the study eye and will be evaluated through Visit 5 (Month 1). If the Low Dose is considered to be safe, the next higher dose will be administered to Cohort 2.

The same enrollment and safety review procedures will be followed for Cohort 2 (Medium Dose DE-120) and Cohort 3 (High Dose DE-120).

ELIGIBILITY:
Main Inclusion Criteria:

* Understand and provide signed written informed consent
* Diagnosis of chronic subretinal or intraretinal fluid secondary to exudative age-related macular degeneration in the study eye
* At least one lesion in the study eye that meets minimal pathology criteria
* Visual acuity of ≤ 55 ETDRS letter (20/80 Snellen equivalent) or worse in the study eye, excluding No Light Perception
* Reasonably clear media and some fixation in the study eye

Main Exclusion Criteria:

Ocular

* Visual acuity of No Light Perception
* Aphakic or has an anterior chamber intraocular lens in the study eye.
* Use or anticipated use of any intravitreal, periocular or photodynamic therapy in the study eye for the treatment of AMD within a specified timeframe prior to Visit 1
* Uncontrolled glaucoma, chronic hypotony or vitrectomy in the study eye
* Evidence of any other ocular disease other than late stage exudative age related macular degeneration in the study eye that may confound the outcome of the study .
* Proscribed ocular surgery in the study eye either prior to or during the course of the trial
* Presence or history of certain ocular or periocular pathology or conditions that could limit ability to perform required study assessments in either eye and/or confound study results

Non-Ocular

* Systemic treatment with anti-VEGF agents (e.g., bevacizumab) is prohibited at any time during the study
* Allergy or hypersensitivity to study drug product, fluorescein dye, or other study related procedures/medications.
* Current or history of certain systemic conditions, abnormalities or therapies that would render a subject a poor candidate for a clinical trial
* Participation in other investigational drug or device clinical trials within 30 days prior to Screening or planning to participate in other investigational drug or device clinical trials for the duration of the study
* Females who are pregnant or lactating and females of child-bearing potential who are not using adequate contraceptive precautions and men who do not agree to practice an acceptable method of contraception throughout the course of the study
* Unable to comply with study procedures or follow-up visits

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04-21 (Actual); Study Completion 2016-04-21 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Each visit from Day 1 to Study Exit (Month 24)
  Adverse events will be assessed at each visit to assess safety
Change from Baseline in central subfield thickness (CST) | Each visit from Day 1 through Study Exit (Month 24)
  CST will be measured using spectral domain optical coherence tomography (SD-OCT)
Change from Baseline in macular volume | Each visit from Day 1 through Study Exit (Month 24)
  Macular volume will be measured using spectral domain optical coherence tomography (SD-OCT)
Drug concentration in plasma over time after a single injection of DE-120 | Most visits from Day 1 through Study Exit (Month 24)
  Pharmacokinetic assessments will include area under the plasma concentration time curve (AUC), peak plasma concentration (Cmax), time to peak plasma concentration (tmax) and elimination half life (t1/2)

SECONDARY OUTCOMES:
Change from Baseline in ocular signs and symptoms | Each visit from Day 1 through Study Exit (Month 24)
  Ocular signs and ocular symptoms will be collected at each visit using slit lamp biomicroscopy, corrected visual acuity, ophthalmoscopy and intraocular pressure measurements

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Bakersfield, California
  - Beverly Hills, California
  - Dallas, Texas